CLINICAL TRIAL: NCT02083861
Title: ZetrOZ Wearable Ultrasound Clinical Study
Brief Title: Wearable LITUS Device for Osteoarthritis of the Knee: a Randomized Double-Blind Placebo-Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OA-03; 1R43MD008597-01 (NIH)
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; arthritis; musculoskeletal; connective tissue disease; ultrasound; pain; mobility; heat; strength; ZetrOZ; LITUS; Sam; grade 1; grade 2
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis; Connective Tissue Diseases; Pain; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active ultrasound device (Experimental): Patients receive treatment from the Sam Ultrasonic Diathermy Device for 4 hours every day for 6 weeks. The active device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Interventions: Device: Sam Ultrasonic Diathermy Device
- Placebo ultrasound device (Placebo Comparator): Patients wear the Sam Ultrasonic Diathermy Device for 4 hours every day for 6 weeks. The placebo device appears and operates identically to the active device except that it does not emit ultrasound.
  Interventions: Device: Sam Ultrasonic Diathermy Device

INTERVENTIONS:
Device: Sam Ultrasonic Diathermy Device — Patients apply the Sam Ultrasonic Diathermy Device daily for 4 hours of continuous therapeutic ultrasound at 3 megahertz (MHz) frequency and 0.132 Watts/cm2.
  Other Names: ZetrOZ ultrasound device; wearable ultrasound device; long duration ultrasound; LITUS device; long duration low intensity device

SUMMARY:
The purpose of this study is to measure the effectiveness of a wearable therapeutic ultrasound device in patients with stage I and stage II knee osteoarthritis. The ability of the device to reduce pain, increase mobility, increase range of motion and muscle strength of the affected leg, and improve quality of life in patients with knee osteoarthritis will be evaluated.

DETAILED DESCRIPTION:
This is an eight week study to clinically evaluate the effect of the low intensity long duration ultrasound (LITUS) device on symptoms of patients suffering from knee osteoarthritis. The device, sam® has been FDA-cleared for use. For the first two weeks of the study, baseline data will be collected as patients report pain scores (NRS) three times per day. During the following 6 weeks, patients will self-apply the wearable LITUS device to their affected knee for 4 hours daily. Each day of the study, pain scores (NRS) will be recorded immediately before application of LITUS device as well as 30 minutes, 2-hours and 4-hours after applying the device. A quality of life assessment (WOMAC), muscle strength and range of motion assessment (JTech) will be performed prior to the patient beginning the protocol and at the conclusion of the protocol.

Up to 93 subjects will be recruited from neighboring communities to the study site. The study is designed to reach a target patient population which includes rural citizens and socioeconomic disadvantaged individuals where non-pharmacotherapies do not exist to manage pain. Subjects will be randomly assigned to active (60%) and placebo groups (40%). The sponsor and investigators are blinded as to which type of device each patient is assigned.

The study will be monitored by an external monitor and a data safety monitoring board (DSMB).

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed mild to moderate knee osteoarthritis (OARSI atlas grades 1-2) based on fixed-flexion x-ray radiological findings for osteophytes and joint space narrowing within the past 12 months
* Fulfill the American College of Rheumatology clinical and radiological diagnostic criteria for knee OA
* 35-80 years of age
* Report a frequent pain score between 3-7 (NRS range: 0-10) during the week preceding enrollment
* Report that knee pain negatively affects quality of life
* Willing not to use any cream, gel, or topical solution during the administration of treatment other than the approved ultrasound gel provided to the subject at the initiation of the study
* Deemed appropriate by their physician or by the study site physician to participate

Exclusion Criteria:

* Cannot successfully demonstrate the ability to put on and take off the device
* Display any condition which, in the judgment of the investigator, would make participation in the study unacceptable, including, but not limited to, the subject's ability to understand and follow instructions.
* Have severe OA or have little to no cartilage in the knee
* Have knee replacement, other surgical intervention, or hyaluronidase injection in the affected knee in the past 6 months
* Are non-ambulatory
* Participated in a clinical trial for an investigational drug and/or agent within 30 days prior to screening
* Modify their medications during the course of the study (medications and doses must remain constant throughout the study)
* Currently taking steroids
* Have contraindication to radiograph
* Have a secondary cause of arthritis (metabolic or inflammatory)

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Ortiz, D.O., MPH, Principal Investigator — Medical Pain Consultants
Locations (1):
- Medical Pain Consultants, Dryden, New York, United States

REFERENCES:
- [Derived] Draper DO, Klyve D, Ortiz R, Best TM. Effect of low-intensity long-duration ultrasound on the symptomatic relief of knee osteoarthritis: a randomized, placebo-controlled double-blind study. J Orthop Surg Res. 2018 Oct 16;13(1):257. doi: 10.1186/s13018-018-0965-0. PMID 30326947

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Ultrasound Device: Patients (n=55) receive treatment from the Sam Ultrasonic Diathermy Device for 4 hours every day for 6 weeks. The active device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Sam Ultrasonic Diathermy Device: Patients apply the Sam Ultrasonic Diathermy Device daily for 4 hours of continuous therapeutic ultrasound at 3 megahertz (MHz) frequency and 0.132 Watts/cm2.
- Placebo Ultrasound Device: Patients (n=35) wear the Sam Ultrasonic Diathermy Device for 4 hours every day for 6 weeks. The placebo device appears and operates identically to the active device except that it does not emit ultrasound.
  Sam Ultrasonic Diathermy Device: Patients apply the Sam Ultrasonic Diathermy Device daily for 4 hours of continuous therapeutic ultrasound at 3 megahertz (MHz) frequency and 0.132 Watts/cm2.
Period: Overall Study
Arm/Group | Active Ultrasound Device | Placebo Ultrasound Device
Started | 57 | 36
Treated | 55 | 35
Completed | 51 | 33
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Ultrasound Device | Placebo Ultrasound Device | Total
Number analyzed (Participants) | 55 | 35 | 90
Age, Continuous [Mean (Full Range); unit: Years] — Population: Only patients that completed study included.
  Years
    number analyzed (Participants) | 51 | 33 | 84
    (all) | 53.6 [35 to 80] | 51.1 [35 to 72] | 52.6 [35 to 80]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only patients that completed study included.
  Participants
    number analyzed (Participants) | 51 | 33 | 84
    Female | 28 | 17 | 45
    Male | 23 | 16 | 39
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: Only patients that completed study included.
  kg/m2
    number analyzed (Participants) | 51 | 33 | 84
    (all) | 34.9 (8.9) | 34.5 (8.3) | 34.7 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Pain on the Numeric Rating Scale (NRS) Change From Baseline to Study Conclusion
Description: The numeric rating scale (NRS) was used to assess change in pain from baseline to study conclusion. NRS range from 0-10 with 0 being no pain and 10 the worst pain possible.
Time Frame: Baseline, Week 6
Population: Patients that completed the entire study were included in analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Ultrasound Device | Placebo Ultrasound Device
Number analyzed (Participants) | 51 | 33
units on a scale | -1.96 [-2.92 to -1.00] | -0.85 [-1.96 to 0.26]

2. Secondary Outcome: Quality of Life (WOMAC) Change From Baseline
Description: WOMAC questionnaire will be utilized (Western Ontario and McMaster Universities Arthritis Index). WOMAC was divided into 3 categories: pain, stiffness, function and total score. The pain category consists of five scores from 0-10, 0 is no pain 10 is worst pain possible for a range of 0 - 50 points. The stiffness category consists of two scores from 0-10, 0 is no stiffness 10 is worst stiffness possible for a range of 0 - 20 points. The function score consists of 17 scores from 0-10, 0 is normal function and 10 is severely limited function, for a range of 0 - 170 points. Categories were multiplied by 10 for analysis. Total score is the sum of pain, stiffness, and function scores (range of 0 - 2400).
Time Frame: Baseline, Week 6
Population: Patients that completed the entire study were included in analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Ultrasound Device | Placebo Ultrasound Device
Number analyzed (Participants) | 51 | 33
units on a scale
  WOMAC Pain Score Change | -107.3 [-147.6 to -66.8] | -60.8 [-100.3 to -21.2]
  WOMAC Stiffness Score Change | -45.0 [-61.1 to -28.9] | -17.1 [-36.0 to -1.9]
  WOMAC Function Score Change | -352.3 [-480.7 to -224.0] | -220.1 [-334.3 to -105.9]
  WOMAC Total Score Change | -504.6 [-683.4 to -325.7] | -311.2 [-473.4 to -148.9]

3. Secondary Outcome: Range of Motion Change From Baseline in Treated Knee
Description: JTech equipment was used to evaluate range of motion range of motion using an inclinometer (www.jtechmedical.com) in flexion and extension of the treated knee. 0 degrees is fully extended and 150 degrees is normal flexion. Positive flexion change indicates improvement in flexion. Negative extension indicates improvement in extension.
Time Frame: Baseline, Week 6
Population: 17 patient subset was assessed for range of motion pilot data.
Measure: Mean (95% Confidence Interval); unit: Degrees
Groups:
- Active Ultrasound Device: Patients (n=9) receive treatment from the Sam Ultrasonic Diathermy Device for 4 hours every day for 6 weeks. The active device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Sam Ultrasonic Diathermy Device: Patients apply the Sam Ultrasonic Diathermy Device daily for 4 hours of continuous therapeutic ultrasound at 3 megahertz (MHz) frequency and 0.132 Watts/cm2.
- Placebo Ultrasound Device: Patients (n=8) wear the Sam Ultrasonic Diathermy Device for 4 hours every day for 6 weeks. The placebo device appears and operates identically to the active device except that it does not emit ultrasound.
  Sam Ultrasonic Diathermy Device: Patients apply the Sam Ultrasonic Diathermy Device daily for 4 hours of continuous therapeutic ultrasound at 3 megahertz (MHz) frequency and 0.132 Watts/cm2.
Arm/Group | Active Ultrasound Device | Placebo Ultrasound Device
Number analyzed (Participants) | 9 | 8
Degrees
  Flexion Change | -6.38 [-40.5 to 27.8] | -2.22 [-29.1 to 24.6]
  Extension Change | -17.75 [-52.5 to 17.0] | -5.56 [-33.2 to 22.1]

4. Secondary Outcome: Muscle Strength Change From Baseline in Treated Knee
Description: Muscle strength in flexion, extension, and rotation were measured using JTECH muscle testing equipment.
Time Frame: Baseline to 6 Weeks
Population: 17 patient subset was assessed for muscle strength pilot data.
Measure: Mean (95% Confidence Interval); unit: Newtons
Arm/Group | Active Ultrasound Device | Placebo Ultrasound Device
Number analyzed (Participants) | 9 | 8
Newtons
  Flexion | 1.34 [-2.22 to 4.89] | 1.01 [-4.06 to 6.08]
  Rotation | 3.21 [0.23 to 6.06] | 0.68 [-3.89 to 5.25]
  Extension | 1.91 [-3.03 to 6.85] | 1.60 [-2.74 to 5.94]

ADVERSE EVENTS:
Time Frame: 8 weeks (study duration)
Description: No adverse events (serious or non-serious) were observed. Patients were supplied with daily diaries where adverse reactions could be self reported. Additionally, follow-up appointments assessed for adverse reactions during weeks 1, 3 (baseline) and week 5, 7, 8 (intervention period).
Arm/Group | Active Ultrasound Device | Placebo Ultrasound Device
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/35
Other Adverse Events (participants affected / at risk) | 0/55 | 0/35

LIMITATIONS AND CAVEATS:
Small number of patients enrolled in range of motion and strength study may have limited statistical analysis. Future studies should include larger sample sizes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No